CLINICAL TRIAL: NCT00852865
Title: Effect of a Dialy Consumption of a Probiotic (Lactobacillus Farciminis) on Hyperalgesia in Response to Thermal Stimulation
Brief Title: Lactobacillus Farciminis and Hyperalgesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lallemand SAS (Industry)
Responsible Party: Henri DURAND, LALLEMAND SAS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HN 08-17; 2008-A01380-55
Record Dates: First submitted 2009-02-25; First posted 2009-02-27 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Inflammation; Pain
Keywords: Inflammation; Pain
MeSH Terms: conditions — Inflammation; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 24 healthy volunteers consuming L.farciminis during three weeks
  Interventions: Drug: Lactobacillus farciminis
- 2 (Placebo Comparator): 24 healthy volunteers consuming placebo during three weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactobacillus farciminis — 1 capsule per day. Each capsule containing 4*109 CFU
  Arms: 1
Drug: Placebo — 1 capsule per day
  Arms: 2

SUMMARY:
We want to analyse a possible effect of o dialy consumption of Lactobacillus farciminis on a hyperalgesia on response to thermal stimulation. A comparaison of results before and after three weeks of treatment will be made.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* consumption of yogurts

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Measurement of the mchanical pain threshold in primary and secondary areas by using a punctate stimulus.

SECONDARY OUTCOMES:
Measurement of cutaneous temperature of hyperalgesia areas

CONTACTS AND LOCATIONS:
Overall Officials: Claude DUBRAY, Professor, Principal Investigator — CPC/CIC-INSERM 501
Locations (1):
- Cpc / Cic-Inserm 501, Clermont-Ferrand, France